CLINICAL TRIAL: NCT05160259
Title: Radial Visualization of the Foramen Arcuale Atlantis
Status: Active, not recruiting | Type: Observational
Sponsor: Samarkand State Medical Institute (Other)
Responsible Party: Sponsor
Other Study IDs: Project#5
Record Dates: First submitted 2021-12-03; First posted 2021-12-16 (Actual); Last update posted 2021-12-16 (Actual); Status verified 2021-12

CONDITIONS: Patients With Kimmerle's Anomaly
Keywords: Kimmerle anomaly, vertebral artery, craniovertebral insufficiency, computed tomography, transcranial Doppler

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Radiation: Radial visualization of the foramen arcuale atlantis — In patients with diagnosed Kimmerle's anomaly, using transcranial Doppler sonography to determine the degree of changes in blood flow in the vertebral arteries

SUMMARY:
Hemodynamics in the craniovertebral zone is often disturbed under the influence of a spondylogenic factor A complication of such changes can be from a slight decrease in cerebral circulation to ischemic changes in the vascular bed The patients underwent complex radiation diagnostics of the craniovertebral region of patients with verified Kimmerle's anomaly (N = 62) All examined patients underwent multispiral computed tomography (CT), ultrasound Doppler and transcranial Doppler (TCD) of the vertebral arteries (VA) Studies of the developmental variant of the first cervical vertebra with the presence of a bony bridge have shown that Kimmerle's anomaly can occur in all age groups

DETAILED DESCRIPTION:
The vaulted hole was found in all age groups (more in young and middle age) The detection rate was within 16 3% of cases, that is, it occurs in every 5-6 people According to TCD data, Kimmerle's anomaly affects blood flow and was most often detected on both sides of the atlas In the unilateral variant, the anomaly was noted only on the left side It was found that the main structural change in the cerebral vascular bed, according to ultrasound diagnostics, is a change in the straightness of the vertebral arteries in the transverse processes of the cervical spine, including the atlas It should also be borne in mind that due to the complexity and mobility of the structure, patients with dysfunction of the craniovertebral zone receive therapy from doctors of various profiles, which requires a comprehensive diagnosis of this problem

ELIGIBILITY:
Inclusion Criteria:

* patients manifested themselves in the form of dizziness, various types of headache, mainly localized in the occipital region, nausea or flashing of flies before the eyes, in the rest - only cervicalgia

Exclusion Criteria:

* acute stroke, brain tumor

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: In patients diagnosed with Kimmerle's anomaly manifested themselves in the form of dizziness, various types of headache, mainly localized in the occipital region, nausea or flashing of flies before the eyes, in the rest - only cervicalgia
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2020-02-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Radial visualization of the foramen arcuale atlantis | up to 36 months
  acute stroke, brain tumor

CONTACTS AND LOCATIONS:
Locations (1):
- Samarkand State Medical Institute, Samarkand, Uzbekistan